CLINICAL TRIAL: NCT01475214
Title: Musculoskeletal Benefits of Bicarbonate in Older Adults - A Dose-Finding Trial
Brief Title: Musculoskeletal Effects of Bicarbonate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Bess Dawson-Hughes, Professor of Medicine, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2705; R01AR060261 (NIH)
Record Dates: First submitted 2011-11-16; First posted 2011-11-21 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Muscle Loss; Fractures; Osteoporosis, Age Related; Fall Injury
Keywords: potassium bicarbonate; urinary N-telopeptide; urinary nitrogen; net acid excretion
MeSH Terms: conditions — Muscular Atrophy; Fractures, Bone; Osteoporosis | interventions — potassium bicarbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- potassium bicarbonate low dose (Active Comparator): potassium bicarbonate in dose of 1.0 mmol/kg per day, given in three even daily doses after meals with a full glass of water
  Interventions: Dietary Supplement: potassium bicarbonate
- potassium bicarbonate higher dose (Active Comparator): potassium bicarbonate in dose of 1.5 mmol/kg per day, given in three even daily doses after meals with a full glass of water
  Interventions: Dietary Supplement: potassium bicarbonate
- placebo (Placebo Comparator): microcrystalline cellulose
  Interventions: Other: Inactive placebo capsule

INTERVENTIONS:
Dietary Supplement: potassium bicarbonate — potassium bicarbonate in dose of 1.0 mmol/kg per day, given in three even daily doses after meals with a full glass of water
  Arms: potassium bicarbonate low dose
Dietary Supplement: potassium bicarbonate — potassium bicarbonate in dose of 1.5 mmol/kg per day, given in three even daily doses after meals with a full glass of water
  Arms: potassium bicarbonate higher dose
Other: Inactive placebo capsule — microcrystalline cellulose
  Arms: placebo

SUMMARY:
With aging, men and women develop a mild and progressive metabolic acidosis. This occurs as a result of declining renal function and ingestion of acid-producing diets. There is extensive evidence that severe metabolic acidosis causes bone and muscle loss, but the impact of the chronic, mild acidosis on bone and muscle in older individuals has not been established. In a recent study, administration of a single dose of bicarbonate daily for 3 months significantly reduced urinary excretion of N-telopeptide (NTX), a marker of bone resorption and urinary nitrogen, a marker of muscle wasting and improved muscle performance in the women but not the men. These and other data support a potential role for bicarbonate as a means of reducing the musculoskeletal declines that lead to extensive morbidity and mortality in the elderly. Before proceeding to a long-term bicarbonate intervention study, however, it is important to identify the dose of bicarbonate most likely to be optimal and to characterize the subjects who benefit most from it. This double blind, placebo controlled, dose-finding study will evaluate the effects of placebo and two doses of bicarbonate on urinary NTX and nitrogen excretion and on lower extremity performance over a 3 month period in 138 men and 138 women, age 60 and older. Changes in urinary excretion of NTX and nitrogen and in selected measures of lower extremity performance will be compared across the three groups. The safety and tolerability of the interventions will also be evaluated. This investigation should provide needed information on the appropriate dosing regimen for men and women and on the study population that should be enrolled in a future bicarbonate intervention trial to assess the long-term effects of this simple, low cost intervention on important clinical outcomes including rates of loss in bone and muscle mass, falls, and fractures.

DETAILED DESCRIPTION:
This dose-finding study will evaluate the effects of placebo and two doses of bicarbonate on urinary NTX and nitrogen excretion and on lower extremity performance over a three month period. The lower dose is similar to the dose shown in our recent trial to be effective. This study is a double blind, randomized, placebo-controlled, parallel-group trial in which 138 healthy men and 138 women, age 60 and older, will take potassium bicarbonate in doses of 1.0 or 1.5 mmol/kg of body weight or placebo daily for three months. Changes in urinary excretion of NTX and nitrogen and in measures of lower extremity performance will be compared across the three groups. The safety and tolerability of the interventions will also be evaluated. This investigation should provide needed information on the appropriate dosing regimen and on the study population that should be enrolled in a future bicarbonate intervention trial to assess the long-term effects of this simple, low cost intervention on important clinical outcomes including rates of loss in bone and muscle mass, falls, and fractures.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* age 60 and older
* community dwelling
* women 1 yr since last menses

Exclusion Criteria:

Medications:

1. Oral glucocorticoids for > 10 days in the last 3 months

   * Cortef (hydrocortisone)
   * Prednisone
2. Parenteral glucocorticoids

   • Decadron (dexamethasone)
3. Osteoporosis medications in the last 6 months

   * Forteo (teriparatide)
   * Calcimar, Miacalcin (calcitonin)
   * Evista (raloxifene)
4. Osteoporosis medications in the last 2 years

   * Fosamax (alendronate)
   * Didronel (etidronate)
   * Aredia (pamidronate)
   * Actonel (risedronate)
   * Reclast (zoledronate)
5. Tamoxifen in the last 6 months
6. Calcium/Parathyroid

   * Rocaltrol (calcitriol)
   * Zemplar (paricalcitol)
   * Drisdol, Ergocalciferol
7. Diuretics currently

   * hydrocholorothiazide (HCTZ)
   * Diuril (chlorothiazide)
   * Thalitone (chlorthalidone)
   * Zaroxolyn (metolazone)
   * Dyazide
   * Maxide
   * Moduretic
   * Lasix (forosamine)
   * Dyrenium (triamterene)
   * Midamor
8. Testosterone or estrogen in the last 6 months (vaginal estrogen okay)
9. Angiotensin converting enzyme (ACE) inhibitors currently

   * Benazepril (Lotensin)
   * Captopril (Capoten)
   * Enalapril (Vasotec)
   * Fosinopril (Monopril)
   * Lisinopril (Prinivil, Zestril)
   * Moexipril (Univasc)
   * Perindopril (Aceon)
   * Quinapril (Accupril)
   * Ramipril (Altace)
   * Trandolapril (Mavik)
10. Angiotensin II receptor blockers currently

    * Candesartan (Atacand)
    * Eprosartan (Teveten)
    * Irbesartan (Avapro)
    * Losartan (Cozaar)
    * Olmesartan (Benicar)
    * Telmisartan (Micardis)
    * Valsartan (Diovan)

Over-the-Counter Drugs currently

1. Antacids - any antacid that contains calcium carbonate, aluminum hydroxide, magnesium hydroxide, or calcium acetate - selected examples include

   * TUMS
   * Mylanta
   * Maalox
   * Titralac
   * Rolaids
   * Sodium bicarbonate (baking soda)
   * Note: magaldrate or Riopan® is allowed
2. Potassium supplements
3. Salt substitutes

Conditions/Diseases

1. renal disease including kidney stones in the past 5 years or glomerular filtration rate (GFR) < 60 ml/min/1.73 m2
2. hyperkalemia (serum potassium >5.3 meq/L; normal range 3.5-5.3 meq/L)
3. elevated serum bicarbonate (serum bicarbonate > 29 mmol/L; normal range 22-29 mmol/L)
4. cirrhosis
5. gastroesophageal reflux disease (GERD) requiring treatment with alkali-containing antacids (TUMS, Mylanta, Maalox, Titralac, Rolaids, or sodium bicarbonate)
6. hyperparathyroidism
7. untreated thyroid disease
8. significant immune disorder such as rheumatoid arthritis
9. current unstable heart disease
10. active malignancy or cancer therapy in the last year
11. fasting spot urine calcium/creatinine > 0.38 mmol/mmol after 1 wk off of calcium supplements
12. congestive heart failure, arrhythmias (surgically treated arrhythmias acceptable), or myocardial infarction in last 12 months
13. serum calcium outside the normal range of 8.3-10.2 mg/dl
14. uncontrolled diabetes mellitus (fasting blood sugar > 130)
15. alcohol use exceeding 2 drinks/day
16. peptic ulcers or esophageal stricture
17. weight <45 or >113.5 kg (<99 or >249.7 lbs)
18. other abnormalities in screening labs, at discretion of the study physician (the PI)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bess Dawson-Hughes, M.D., Principal Investigator — Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Shea MK, Dawson-Hughes B. Association of Urinary Citrate With Acid-Base Status, Bone Resorption, and Calcium Excretion in Older Men and Women. J Clin Endocrinol Metab. 2018 Feb 1;103(2):452-459. doi: 10.1210/jc.2017-01778. PMID 29211866
- [Derived] Ceglia L, Dawson-Hughes B. Increasing alkali supplementation decreases urinary nitrogen excretion when adjusted for same day nitrogen intake. Osteoporos Int. 2017 Dec;28(12):3355-3359. doi: 10.1007/s00198-017-4196-8. Epub 2017 Aug 25. PMID 28842733

RESULTS

PARTICIPANT FLOW:
Groups:
- Inactive Capsule: microcrystalline cellulose
  placebo: microcrystalline cellulose
Period: Overall Study
Arm/Group | Potassium Bicarbonate Low Dose | Potassium Bicarbonate Higher Dose | Inactive Capsule
Started | 84 | 79 | 81
Completed | 79 | 75 | 79
Not Completed | 5 | 4 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Inactive Placebo Capsule: microcrystalline cellulose
  placebo: microcrystalline cellulose
- Total: Total of all reporting groups
Arm/Group | Potassium Bicarbonate Low Dose | Potassium Bicarbonate Higher Dose | Inactive Placebo Capsule | Total
Number analyzed (Participants) | 84 | 79 | 81 | 244
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 41 | 121
  >=65 years | 44 | 39 | 40 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (5.5) | 66.4 (5.1) | 66.8 (6.1) | 66.9 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 39 | 38 | 118
  Male | 43 | 40 | 43 | 126
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian, Non-hispanic | 76 | 68 | 75 | 219
  Caucasian, Hispanic | 2 | 1 | 2 | 5
  African-American | 6 | 9 | 3 | 18
  Asian | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 84 | 79 | 81 | 244
Weight [Mean (Standard Deviation); unit: kg] | 74.8 (13.7) | 74.2 (13.0) | 73.2 (14.0) | 74.1 (13.6)
Glomerular Filtration Rate (GFR) [Mean (Standard Deviation); unit: ml/min/1.73m^2] | 76.5 (13.2) | 77.5 (12.8) | 74.8 (12.9) | 76.3 (13.0)
Serum potassium [Mean (Standard Deviation); unit: meq/L] | 4.31 (0.29) | 4.39 (0.36) | 4.30 (0.31) | 4.33 (0.32)
Serum bicarbonate [Mean (Standard Deviation); unit: mmol/L] | 26.1 (1.9) | 25.8 (2.4) | 26.1 (2.4) | 26.0 (2.2)
Urine calcium/creatinine [Mean (Standard Deviation); unit: mg/g] | 99 (43) | 99 (48) | 114 (69) | 104 (55)

OUTCOME MEASURES:

1. Primary Outcome: The Dose of Potassium Bicarbonate Needed for Maximal Suppression of 24-hr Urinary N-telopeptide
Description: Describe and compare changes in urinary N-telopeptide (NTX) across the placebo and Potassium Bicarbonate (KHCO3) doses.
Time Frame: 84 days
Population: Healthy men and women age 60 years and older
Measure: Mean (Standard Error); unit: nmol/day
Arm/Group | Potassium Bicarbonate Low Dose | Potassium Bicarbonate Higher Dose | Inactive Placebo Capsule
Number analyzed (Participants) | 79 | 75 | 79
nmol/day
  baseline 24-hr urinary NTX | 240 (17) | 230 (20) | 241 (17)
  change in NTX | -53 (11) | -43 (11) | -14 (11)

2. Primary Outcome: Co-primary Aim - to Identify the Dose of KHCO3 Needed for Maximal Suppression of 24-hr Urinary Nitrogen
Description: Describe and compare changes in 24-hour urinary nitrogen in the low and high dose and KHCO3 group and in placebo.
Time Frame: 84 days
Population: healthy men and women age 60 years and older
Measure: Mean (Standard Error); unit: mmol/day
Arm/Group | Potassium Bicarbonate Low Dose | Potassium Bicarbonate Higher Dose | Inactive Capsule
Number analyzed (Participants) | 79 | 75 | 79
mmol/day
  baseline 24-hr urine nitrogen | 769 (32) | 834 (39) | 864 (33)
  change in 24-hr urine nitrogen | -29.4 (18.6) | -16.4 (19.1) | -21.0 (18.7)

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | Potassium Bicarbonate Low Dose | Potassium Bicarbonate Higher Dose | Inactive Capsule
Serious Adverse Events (participants affected / at risk) | 3/84 | 3/79 | 1/81
Other Adverse Events (participants affected / at risk) | 19/84 | 29/79 | 23/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Potassium Bicarbonate Low Dose (N=84) | Potassium Bicarbonate Higher Dose (N=79) | Inactive Capsule (N=81)
High serum potassium (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Contusions/abrasions (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) — Resulting from falls
GI upset (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Bloating, dizziness
Abdominal aortic repair (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Fracture, right wrist, from fall
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Potassium Bicarbonate Low Dose (N=84) | Potassium Bicarbonate Higher Dose (N=79) | Inactive Capsule (N=81)
High serum potassium (Renal and urinary disorders) | 5 (7) | 8 (10) | 5 (9) — Potassium level > 5.3 meq/L
low GFR (Renal and urinary disorders) | 4 (5) | 3 (3) | 3 (3) — Reported if GFR < 55; protocol change GFR < 45
GI upset (Gastrointestinal disorders) | 5 (5) | 9 (11) | 6 (6) — GI upset, heartburn, gas, bloating, nausea
Headache (General disorders) | 1 (1) | 1 (1) | 2 (2) — Headache, migraine
Heart palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Fever, fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
dizziness (General disorders) | 1 (1) | 2 (2) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Knee/hip injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) — Sprain
Sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Mouth irritation (General disorders) | 0 (0) | 0 (0) | 1 (1) — Roof of mouth irritation
Constipation/diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Numbness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Reports numbness in thumb
Skin cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No